CLINICAL TRIAL: NCT04844918
Title: Efficacy and Safety of Once-Weekly Tirzepatide in Participants With Obesity Disease: A Randomized, Double-Blind, Placebo-Controlled Trial (SURMOUNT-J)
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Obesity Disease
Acronym: SURMOUNT-J
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17506; I8F-JE-GPHZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-04-01; First posted 2021-04-14 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Obesity
Keywords: Metabolism and Nutrition Disorder; Obesity Related Health Problems; Obesity Disease
MeSH Terms: conditions — Obesity; Nutrition Disorders | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 10 Milligrams (mg) Tirzepatide (Experimental): Participants received maintenance dose 10 mg with dose escalation starting from 2.5 mg, 5 mg, 7.5 mg and then 10 mg tirzepatide administered subcutaneously (SC) once weekly (QW).
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): Participants received maintenance dose 15 mg with dose escalation starting from 2.5 mg, 5 mg, 7.5 mg, 10 mg, 12.5 mg and then 15 mg tirzepatide administered SC QW.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants received matching placebo administered SC QW.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 Milligrams (mg) Tirzepatide; 15 mg Tirzepatide
Other: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn more about tirzepatide in participants with obesity disease. The study will also measure how Tirzepatide affects body weight with a low-calorie diet and increased physical activity. The study will last around 72 Weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI of greater than or equal to ≥27 kg/m² and <less than 35 kg/m² with at least 2 obesity-related health problems or ≥35 kg/m² with at least 1 obesity-related health problems. Health problems are IGT, hyperlipidemia, or NAFLD.
* Have a history of at least 1 self-reported unsuccessful dietary effort to lose body weight.

Exclusion Criteria:

* Have diabetes.
* Acute or chronic liver disease other than NAFLD.
* Have a self-reported change in body weight >5 kg within 3 months prior to screening.
* Have or plan to have endoscopic and/or device-based therapy for obesity or have had device removal within the last 6 months.
* Have renal impairment measured as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2, calculated by Japanese Society of Nephrology coefficient-modified Chronic Kidney Disease-Epidemiology equation during screening.
* Have a known clinically significant gastric emptying abnormality.
* Have had a history of chronic or acute pancreatitis.
* Have thyroid-stimulating hormone outside of the range of 0.4 to 6.0 micro units per milliliter (μIU/mL) at screening.
* Have obesity induced by other endocrinologic disorders or diagnosed monogenetic or syndromic forms of obesity.
* Have a history of significant active or unstable major depressive disorder or other severe psychiatric disorder within the last 2 years.
* Have a cardiovascular condition within 3 months prior to randomization
* Have a family or personal history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia Syndrome type 2.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLilly (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (18):
- Japan (18):
  - Kohnodai Hospital, National Center for Global Health and Medicine, Ichikawa, Chiba
  - Saiseikai Matsuyama Hospital, Matsuyama, Ehime
  - Takai Internal Medicine Clinic, Kamakura-shi, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Motomachi Takatsuka Naika Clinic, Yokohama, Kanagawa
  - Osaka Saiseikai Suita hospital, Suita, Osaka
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - The Institute for Adult Disease, Asahi Life Foundation, Chuo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Saiseikai Central Hospital, Minato-Ku, Tokyo
  - Shimokitazawa Tomo Clinic, Setagaya-ku, Tokyo
  - Miho Clinic, Shinagawa-ku, Tokyo
  - Medical Corporation Heishinkai ToCROM Clinic, Shinjuku-ku, Tokyo
  - Yamagata Tokushukai Hospital, Yamagata, Yamagata
  - AMC Nishiumeda Clinic, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Yokote K, Fukushima Y, Shingaki T, Oura T, Ogawa W. Association of baseline characteristics with clinical outcomes of tirzepatide treatment in Japanese patients with obesity disease: A subgroup analysis of the SURMOUNT-J trial. Diabetes Obes Metab. 2026 Feb;28(2):1278-1287. doi: 10.1111/dom.70315. Epub 2025 Nov 25. PMID 41290555
- [Derived] Kadowaki T, Kiyosue A, Shingaki T, Oura T, Yokote K. Efficacy and safety of once-weekly tirzepatide in Japanese patients with obesity disease (SURMOUNT-J): a multicentre, randomised, double-blind, placebo-controlled phase 3 trial. Lancet Diabetes Endocrinol. 2025 May;13(5):384-396. doi: 10.1016/S2213-8587(24)00377-2. Epub 2025 Feb 28. PMID 40031941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 267 participants were randomized in the study. However, due to good clinical practice (GCP) compliance issues identified at one of the investigative sites, all 42 participants from that site were excluded from the study analyses
Period: Overall Study
Arm/Group | 10 Milligrams (mg) Tirzepatide | 15 mg Tirzepatide | Placebo
Started | 88 | 90 | 89
Received At Least 1 Dose of Study Drug (Excluding the GCP Compliance Investigative Site) | 73 | 77 | 75
Completed | 60 | 65 | 67
Not Completed | 28 | 25 | 22
Not completed — Adverse Event | 7 | 8 | 5
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 3 | 3
Not completed — Participants Excluded Due to GCP Compliance Issue | 15 | 13 | 14

BASELINE CHARACTERISTICS:
Population: All participants, excluding the GCP compliance investigative site, who received at least one dose of study drug.
Groups:
- 10 mg Tirzepatide: Participants received maintenance dose 10 mg with dose escalation starting from 2.5 mg, 5 mg, 7.5 mg and then 10 mg tirzepatide administered SC QW.
- Total: Total of all reporting groups
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo | Total
Number analyzed (Participants) | 73 | 77 | 75 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.00 (10.87) | 51.10 (10.30) | 52.30 (10.93) | 50.80 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 30 | 92
  Male | 43 | 45 | 45 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 73 | 77 | 75 | 225
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 73 | 77 | 75 | 225
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 73 | 77 | 75 | 225

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Body Weight
Description: Mean percent change in body weight was measured. Least squares (LS) mean was determined using mixed model repeated measures (MMRM) model with Baseline + impaired glucose tolerance (IGT) at Screening + Hyperlipidemia at Screening + non-alcoholic fatty liver disease (NAFLD) at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, 72 Weeks
Population: All participants, excluding the GCP compliance investigative site, who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 59 | 65 | 66
Percent change | -17.8 (0.94) | -22.7 (0.90) | -1.7 (0.90)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -16.1, 95% CI 2-sided [-18.7 to -13.5]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -21.1, 95% CI 2-sided [-23.6 to -18.5]

2. Primary Outcome: Percentage of Participants Who Achieve ≥5% Body Weight Reduction
Description: Percentage of Participants Who Achieve ≥5% Body Weight Reduction
Time Frame: Week 72
Population: All participants, excluding the GCP compliance investigative site, who received at least one dose of study drug, had a baseline and at least one post-baseline value for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 71 | 76 | 75
Percentage of participants | 94.37 | 96.05 | 20
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 119.65, 95% CI 2-sided [29.06 to 492.67]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 153.57, 95% CI 2-sided [36.03 to 654.53]

3. Secondary Outcome: Percentage of Participants Who Had Improvement in Obesity-related Health Problems
Description: Percentage of participants who had improvement in obesity-related health problems
Time Frame: Week 72
Population: All participants, excluding the GCP compliance investigative site, who received at least one dose of study drug and evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 60 | 64 | 63
Percentage of participants | 70.0 | 79.69 | 11.11
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 24.26, 95% CI 2-sided [8.62 to 68.28]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 38.27, 95% CI 2-sided [13.21 to 110.89]

4. Secondary Outcome: Change From Baseline in Fasting Glucose for Participants With IGT at Baseline
Description: Change from Baseline in Fasting Glucose for Participants with IGT at Baseline. LS mean was determined by MMRM model with = Baseline + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: All participants, excluding the GCP compliance investigative site, who had IGT at baseline, received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 35 | 40 | 47
milligrams per deciliter (mg/dL) | -12.81 (1.490) | -10.61 (1.391) | 2.19 (1.291)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -15.00, 95% CI 2-sided [-18.91 to -11.09]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -12.80, 95% CI 2-sided [-16.56 to -9.05]

5. Secondary Outcome: Change From Baseline in Oral Glucose Tolerance (OGTT) 2-hr Glucose for Participants With Impaired Glucose Tolerance (IGT) at Baseline
Description: Change from Baseline in OGTT 2-hr Glucose for Participants with IGT at Baseline. LS mean was determined by MMRM model with Baseline + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 35 | 40 | 47
milligrams per deciliter (mg/dL) | -61.50 (5.330) | -70.56 (4.951) | -5.74 (4.612)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -55.76, 95% CI 2-sided [-69.74 to -41.77]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -64.82, 95% CI 2-sided [-78.20 to -51.43]

6. Secondary Outcome: Percent Change From Baseline in Fasting Lipids [Triglycerides (TG)] for Participants With Hyperlipidemia at Baseline
Description: Percent Change from Baseline in Fasting Lipids TG for Participants with Hyperlipidemia at Baseline. LS mean was determined by MMRM model with log (Baseline) + NAFLD at Screening + IGT at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: All participants, excluding the GCP compliance investigative site, who had hyperlipidemia at baseline, received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 29 | 37 | 36
Percent change | -47.3 (3.34) | -50.6 (2.77) | -11.0 (5.14)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -40.7, 95% CI 2-sided [-50.0 to -29.7]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -44.5, 95% CI 2-sided [-52.7 to -34.9]

7. Secondary Outcome: Percent Change From Baseline in Hepatic Fat Fraction (HFF) for Participants With Non-alcoholic Fatty Liver Disease [NAFLD]
Description: Percent Change from Baseline in HFF for participants diagnosed as NAFLD by MRI at Baseline. LS mean was determined by ANCOVA model with Baseline + Hyperlipidemia at Screening + IGT at Screening + Sex + Treatment (Type III sum of squares) as variables. Percent Change from Baseline in HFF for participants with NAFLD is reported. NAFLD was diagnosed by Magnetic Resonance Imaging (MRI) at Baseline. This was evaluated only for participants who were diagnosed with NAFLD at baseline by MRI.
Time Frame: Baseline, Week 72
Population: All participants, excluding the GCP compliance investigative site, who were diagnosed as NAFLD by MRI at baseline and received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 59 | 62 | 61
Percent change | -63.9 (3.09) | -69.9 (2.99) | -19.6 (3.05)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -44.4, 95% CI 2-sided [-53.0 to -35.7]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -50.4, 95% CI 2-sided [-58.8 to -41.9]

8. Secondary Outcome: Percentage of Participants Who Achieved Improvements of IGT
Description: Percentage of Participants Who Achieved Improvements of IGT. This was evaluated only for participants with IGT at baseline.
Time Frame: Week 72
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 40 | 46 | 50
Percentage of participants | 92.50 | 97.83 | 28.0
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 25.42, 95% CI 2-sided [7.25 to 89.14]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 70.66, 95% CI 2-sided [12.73 to 392.24]

9. Secondary Outcome: Percentage of Participants Who Achieved Improvements of Hyperlipidemia
Description: Percentage of Participants Who Achieved Improvements of Hyperlipidemia. This was evaluated only for participants with hyperlipidemia at baseline.
Time Frame: Week 72
Population: All participants, excluding the GCP compliance investigative site, with hyperlipidemia at baseline, received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 29 | 37 | 36
Percentage of participants | 72.41 | 81.08 | 25
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 9.29, 95% CI 2-sided [2.86 to 30.20]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 15.67, 95% CI 2-sided [4.78 to 51.37]

10. Secondary Outcome: Percentage of Participants Who Achieved Improvements of NAFLD
Description: Percentage of Participants Who Achieved Improvements of NAFLD. This was evaluated only for participants who were diagnosed as NAFLD by MRI at Baseline.
Time Frame: Week 72
Population: All participants, excluding the GCP compliance investigative site, diagnosed as NAFLD by MRI at baseline, received at least one dose of study drug, and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 59 | 62 | 61
Percentage of participants | 69.49 | 77.42 | 9.84
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 27.50, 95% CI 2-sided [9.35 to 80.88]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 40.01, 95% CI 2-sided [13.27 to 120.57]

11. Secondary Outcome: Percentage of Participants Who Achieve ≥10% Body Weight Reduction
Description: Percentage of Participants Who Achieve ≥10% body weight reduction.
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 71 | 76 | 75
Percentage of participants | 85.92 | 92.11 | 4
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 185.92, 95% CI 2-sided [46.39 to 745.16]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 318.02, 95% CI 2-sided [74.49 to 1357.79]

12. Secondary Outcome: Percentage of Participants Who Achieve ≥15% Body Weight Reduction
Description: Percentage of Participants Who Achieve ≥15% body weight reduction.
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 71 | 76 | 75
Percentage of participants | 63.38 | 82.89 | 1.33
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 100.21, 95% CI 2-sided [18.64 to 538.74]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 286.73, 95% CI 2-sided [50.68 to 1622.06]

13. Secondary Outcome: Change From Baseline in Absolute Body Weight
Description: Change from Baseline in Absolute Body Weight. LS mean was determined by MMRM model with Baseline + IGT at Screening + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 59 | 65 | 66
kilograms (kg) | -16.0 (0.86) | -20.8 (0.82) | -1.5 (0.82)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -14.5, 95% CI 2-sided [-16.8 to -12.2]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -19.3, 95% CI 2-sided [-21.6 to -17.0]

14. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Change from Baseline in BMI. LS mean was determined using MMRM model with Baseline + IGT at Screening + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms per metres squared (kg/m^2)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 59 | 65 | 66
kilograms per metres squared (kg/m^2) | -5.8 (0.32) | -7.7 (0.30) | -0.6 (0.30)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -5.2, 95% CI 2-sided [-6.1 to -4.4]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -7.1, 95% CI 2-sided [-8.0 to -6.3]

15. Secondary Outcome: Percent Change From Baseline in Visceral Adipose Tissue (VAT)
Description: Percent Change from Baseline in VAT. LS mean was determined by MMRM model with Baseline + IGT at Screening + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 60 | 63 | 61
Percent change | -39.4 (2.44) | -44.5 (2.37) | -3.4 (2.42)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -36.1, 95% CI 2-sided [-42.9 to -29.3]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -41.1, 95% CI 2-sided [-47.8 to -34.4]

16. Secondary Outcome: Percent Change From Baseline in Subcutaneous Adipose Tissue (SAT)
Description: Percent Change from Baseline in SAT. LS mean was determined by MMRM model with Baseline + IGT at Screening + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 60 | 63 | 61
Percent change | -32.2 (1.90) | -36.5 (1.85) | -5.0 (1.90)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -27.2, 95% CI 2-sided [-32.6 to -21.9]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -31.5, 95% CI 2-sided [-36.7 to -26.2]

17. Secondary Outcome: Change From Baseline in VAT/SAT Ratio
Description: Change from Baseline in VAT/SAT Ratio. LS mean was determined by MMRM model with Baseline + IGT at Screening + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 60 | 63 | 61
ratio | -0.09 (0.023) | -0.08 (0.023) | 0.01 (0.023)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.004, Mixed Models Analysis; LS Mean Difference = -0.10, 95% CI 2-sided [-0.16 to -0.03]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.006, Mixed Models Analysis; LS Mean Difference = -0.09, 95% CI 2-sided [-0.15 to -0.03]

18. Secondary Outcome: Percentage of Participants Who Achieved VAT <100 Square Centimeter (cm²) From Baseline for Participants With VAT≥100 cm² at Baseline
Description: Percentage of Participants Who Achieve VAT <100 cm² from Baseline for participants with VAT≥100 cm² at Baseline.
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 57 | 62 | 61
Percentage of participants | 26.32 | 37.10 | 1.64
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 28.52, 95% CI 2-sided [4.31 to 188.55]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 57.73, 95% CI 2-sided [8.68 to 383.88]

19. Secondary Outcome: Change From Baseline in Waist Circumference
Description: Change from Baseline in Waist Circumference. LS mean was determined using MMRM model with = Baseline + IGT at Screening + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: centimeters (cm)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 59 | 65 | 66
centimeters (cm) | -12.7 (0.88) | -16.6 (0.83) | -1.3 (0.84)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -11.4, 95% CI 2-sided [-13.8 to -9.0]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -15.3, 95% CI 2-sided [-17.7 to -13.0]

20. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: Change from Baseline in HbA1c was assessed only for Participants with IGT at Baseline. LS mean was determined using MMRM model with = Baseline + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 35 | 40 | 47
Percentage of HbA1c | -0.67 (0.045) | -0.68 (0.042) | -0.02 (0.039)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.65, 95% CI 2-sided [-0.77 to -0.53]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.66, 95% CI 2-sided [-0.77 to -0.55]

21. Secondary Outcome: Change From Baseline in Fasting Insulin for Participants With IGT at Baseline
Description: Change from Baseline in Fasting Insulin for Participants with IGT at Baseline. LS mean was determined using MMRM model log(Baseline) + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: All participants, excluding the GCP compliance investigative site, who had IGT at baseline, received at least one dose of study drug, and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: milli-international units/liter (mIU/L)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 34 | 37 | 46
milli-international units/liter (mIU/L) | -6.04 (0.517) | -6.69 (0.433) | -2.13 (0.776)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; LS Mean Difference = -3.91, 95% CI 2-sided [-5.74 to -2.08]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; LS Mean Difference = -4.55, 95% CI 2-sided [-6.29 to -2.81]

22. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Description: Change from Baseline in Systolic Blood Pressure. LS mean was determined using MMRM model with Baseline + Hyperlipidemia at Screening + NAFLD at Screening + IGT at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeters of Mercury (mmHg)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 59 | 65 | 66
millimeters of Mercury (mmHg) | -11.2 (1.42) | -12.0 (1.35) | 1.9 (1.35)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -13.2, 95% CI 2-sided [-17.0 to -9.3]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -13.9, 95% CI 2-sided [-17.7 to -10.1]

23. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: Change from Baseline in Diastolic Blood Pressure. LS mean was determined using MMRM model with Baseline + Hyperlipidemia at Screening + NAFLD at Screening + IGT at Screening + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeters of Mercury (mmHg)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 59 | 65 | 66
millimeters of Mercury (mmHg) | -5.9 (1.09) | -6.3 (1.04) | 0.5 (1.04)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -6.3, 95% CI 2-sided [-9.3 to -3.4]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -6.8, 95% CI 2-sided [-9.7 to -3.9]

24. Secondary Outcome: Change From Baseline in Short Form 36 Version 2 Health Survey (SF-36v2) Acute Form Physical Functioning Domain Score
Description: The SF-36v2 acute form, 1-week recall assesses participants' health-related quality of life (HRQoL) on 8 domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Information from these 8 domains is further aggregated into 2 health component summary scores: Physical Component Summary and Mental Component Summary.
  Items are answered on Likert scales of varying lengths. Scoring of each domain and both summary scores are norm based and presented in the form of T scores, with a mean of 50 and standard deviation of 10; higher scores indicate better levels of function and/or better health. Range cannot be specified in norm-based scores. LS mean was determined using ANCOVA model with Week 0 (Visit 3) + IGT at Screening + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 63 | 68 | 69
Score on a scale | 1.1 (0.39) | 2.0 (0.37) | -0.1 (0.37)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.022, ANCOVA; LS Mean Difference = 1.3, 95% CI 2-sided [0.2 to 2.3]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 2.1, 95% CI 2-sided [1.1 to 3.2]

25. Secondary Outcome: Change From Baseline in Impact of Weight on Quality-of-Life Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function Composite Score
Description: The IWQOL Lite-CT consists of 20 items, assessing 2 primary domains of obesity related HRQoL: Physical (7 items) and Psychosocial (13 items). A 5-item subset of the Physical domain - the Physical Function composite - is also supported. Items in the Physical Function composite describe physical impacts related to general and specific physical activities. All items in the physical domain are rated on either a 5-point frequency ("never" to "always") scale or a 5-point truth ("not at all true" to "completely true") scale. Total score of IWQOL-Lite-CT composite ranges from 0 to 100, with higher scores reflecting better quality of life. LS mean was determined using ANCOVA model with Week 0 (Visit 3) + IGT at Screening + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 63 | 69 | 69
Score on a scale | 15.2 (2.05) | 13.0 (1.95) | 2.2 (1.96)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 13.0, 95% CI 2-sided [7.4 to 18.7]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 10.8, 95% CI 2-sided [5.4 to 16.3]

26. Secondary Outcome: Change From Baseline in Euro Quality of Life Five Dimensions (EQ-5D-5L)
Description: The EQ-5D-5L is a standardized instrument used to measure self-reported health status of the participants. It comprises of 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). There are 5 response levels (no problems, slight problems, moderate problems, severe problems, unable to perform/extreme problems). In addition to the health profile, a single health state index value can be derived based on a formula that attaches weights to each of the levels in each dimension. This index value ranges between
  ˂0 (where 0 is a health state equivalent to death; negative values are valued as worse than dead) to 1 (perfect health). LS mean was determined using ANCOVA model with Week 0 (Visit 3) + IGT at Screening + Hyperlipidemia at Screening + NAFLD at Screening + Sex + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 63 | 68 | 69
Score on a scale | 0.01 (0.011) | 0.01 (0.011) | -0.01 (0.011)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.099, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [0.00 to 0.06]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.236, ANCOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.01 to 0.05]

ADVERSE EVENTS:
Time Frame: Baseline Through Safety Follow-Up (Up To 76 Weeks)
Description: All participants, excluding the GCP compliance investigative site, who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly. Based on the planned safety analysis, adverse events were collected per the treatment regimen, irrespective of each dose level.
Groups:
- 10 mg Tirzepatide: Participants received maintenance dose 10 mg with dose escalation starting from 2.5 mg, 5 mg, 7.5 mg and then 10 mg tirzepatide SC QW
  .
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/77 | 0/75
Serious Adverse Events (participants affected / at risk) | 8/73 | 5/77 | 5/75
Other Adverse Events (participants affected / at risk) | 59/73 | 65/77 | 51/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 10 mg Tirzepatide (N=73) | 15 mg Tirzepatide (N=77) | Placebo (N=75)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/30 (0) | 1/32 (1) | 0/30 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/43 (1) | 0/45 (0) | 0/45 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/30 (0) | 1/32 (1) | 0/30 (0)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/43 (0) | 0/45 (0) | 1/45 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 10 mg Tirzepatide (N=73) | 15 mg Tirzepatide (N=77) | Placebo (N=75)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Conductive deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 1 (2)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 5 (11) | 4 (6) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 12 (14) | 21 (23) | 5 (16)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 9 (15) | 7 (8) | 3 (3)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (6) | 3 (3) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (31) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (13) | 18 (40) | 3 (3)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (11) | 9 (11) | 3 (3)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (8) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 4 (43) | 4 (28) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (5) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 10 (10) | 11 (15) | 11 (14)
Vaccination site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vaccination site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 2 (3)
Bartholin's abscess (Infections and infestations) | 1/30 (1) | 0/32 (0) | 0/30 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 15 (15) | 15 (15) | 13 (14)
Cystitis (Infections and infestations) | 0 (0) | 3 (5) | 1 (1)
Folliculitis genital (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (4) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (11) | 1 (1) | 8 (9)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea manuum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (2) | 4 (4) | 4 (4)
Post vaccination fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Albumin urine present (Investigations) | 0 (0) | 0 (0) | 3 (3)
Amylase increased (Investigations) | 3 (3) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood calcitonin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Helicobacter test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1/43 (1) | 0/45 (0) | 0/45 (0)
Protein urine present (Investigations) | 1 (1) | 2 (2) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 6 (7) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3) | 4 (6)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal submucosal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/30 (0) | 1/32 (1) | 0/30 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (4) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 5 (6)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0/30 (0) | 0/32 (0) | 1/30 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 0/30 (0) | 1/32 (1) | 0/30 (0)
Prostatitis (Reproductive system and breast disorders) | 1/43 (1) | 0/45 (0) | 0/45 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord atrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Mass excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 0/43 (0) | 0/45 (0) | 1/45 (1)
Artery dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT04844918/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT04844918/SAP_001.pdf